CLINICAL TRIAL: NCT05412134
Title: Inspiratory Muscle Rehabilitation in Children With Obesity to Promote Physical Activity
Brief Title: Inspiratory Muscle Rehabilitation in Children With Obesity
Acronym: BREATHE Fit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: The Derfner Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00110494
Record Dates: First submitted 2022-06-07; First posted 2022-06-09 (Actual); Results first posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Pediatric Obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The only person who will know the arm of each participant will be the study team member in charge of randomization (the clinical research coordinator)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active inspiratory muscle rehabilitation (IMR) group (Experimental): Each participant will be provided a PrO2™ device and trained on its use and its accompanying PrO2 Fit™ app. The PrO2™ is a flow-resistive device that provides inspiratory resistance via a fixed 2mm orifice and has Bluetooth connectivity to most IOS/Android devices or Mac/Windows computers. The PrO2™ device and app allows for both 100% adherence monitoring and immediate user biofeedback.
  Participants will be instructed at Visit 1 and Visit 2 to inspire forcefully through PrO2™ until the device signals that the user has achieved the target resistance (via audible alarm and visible light signal). The research team will implement biofeedback signals at a specific inspiratory resistance to provide a precise and individualized training target. Successful IMR repetitions will require that subjects achieve a pressure target that is 75% of their MIP.
  Interventions: Device: Pro2 - 75% of participant's MIP
- SHAM (Active Comparator): Participants in the control intervention will also use the same PrO2™ device but at a reduced peak resistance of 15% MIP. The research team will implement biofeedback signals at a specific inspiratory resistance to provide precise and individualized training target. Successful IMR repetitions will require that subjects achieve a pressure target that is 15% of their MIP for each repetition. Participants will perform 3 sets of 50 inspiratory breaths 3 times per week.
  Interventions: Device: Pro2 - 15% of participant's MIP

INTERVENTIONS:
Device: Pro2 - 75% of participant's MIP — Each participant will be provided a PrO2™ device and trained on its use as well as its accompanying PrO2 Fit™ app. The PrO2™ is a flow-resistive device that provides inspiratory resistance via a fixed 2mm orifice and has Bluetooth connectivity to most IOS/Android devices or Mac/Windows computers. The PrO2™ device and app allows for both 100% adherence monitoring and immediate user biofeedback.
  Participants will be instructed to inspire forcefully through PrO2™ until the device signals that the user has achieved the target resistance (via audible alarm and visible light signal). The research team will implement biofeedback signals at a specific inspiratory resistance to provide precise and individualized training target. Successful IMR repetitions will require that subjects achieve a pressure target that is 75% of their MIP.
  Arms: Active inspiratory muscle rehabilitation (IMR) group
Device: Pro2 - 15% of participant's MIP — Participants in the control intervention will also use the same PrO2™ device but at a reduced peak resistance of 15% MIP. The research team will implement biofeedback signals at a specific inspiratory resistance to provide precise and individualized training target. Successful IMR repetitions will require that subjects achieve a pressure target that is 15% of their MIP for each repetition. Participants will perform 3 sets of 50 inspiratory breaths 3 times per week.
  Arms: SHAM

SUMMARY:
This is a single-center, randomized, SHAM-controlled, parallel assignment, double-masked, interventional trial among children aged 8-17 years (not yet 18 years old) of age with obesity (n=30), recruited from the Duke Healthy Lifestyles Clinic to test the effectiveness of inspiratory muscle rehabilitation (IMR) as an acceptable add-on intervention to reduce dyspnea (feeling short-of-breath or breathless) and to promote greater activity in children with obesity

DETAILED DESCRIPTION:
Improved management of obesity is an urgent public health need. Nearly 40% of US children and adolescents have a body mass index that markedly increases their risk for serious metabolic and cardiopulmonary sequelae. Current childhood obesity rates, for the first time in US history, predict a decline in life US expectancy. Importantly, childhood obesity is a key driver of health disparities in the US, with obesity disproportionately affecting African-American, Hispanic-Latino, and Native American children. A key contributor to the sequelae of obesity is sedentariness. Thus, best practice in obesity management includes both reducing sedentariness and establishing durable increases in daily physical activity, however, attrition from planned exercise programs remains high. A key challenge to initiating and sustaining physical activity in children with obesity is the extreme dyspnea (breathlessness) they experience. This is due to the altered thoracic mechanics of obesity which lead to enhanced inspiratory muscle fatigue and dyspnea, with even modest physical activity. Our group has confirmed that among adolescents, higher body mass index (BMI) associates with lower inspiratory muscle endurance (r= -0.680, p=0.049, n=14), and that this lower endurance correlates with more frequent dyspnea (r= - 0.672, p=0.023, n=12). Treating obesity-related inspiratory muscle impairment and dyspnea is a promising approach to support physical activity in children with obesity but is yet unproven.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent from legal guardian and assent from participant as appropriate.
* Children 8 to 17 years of age with obesity (BMI ≥ 95th percentile for age and sex) being seen at Duke Healthy Lifestyles clinic.
* Participants (or parent/guardian) must have access to the internet and an approved smart device/computer.
* Child must have a designated caregiver who expresses a commitment to encourage the participant to complete the study procedures.
* Participant and legal guardian must speak and read English.

Exclusion Criteria:

* Prior enrollment in an IMR program.
* Contraindications for IMR including a history of recent lung surgery, recent pulmonary embolism, or history of recurrent spontaneous pneumothorax
* Progressive neurological or neuromuscular disorders or need for chronic O2 therapy.
* Inability to complete baseline measurements in a satisfactory manner according to the judgment of the research coordinator or PI.
* Current self-reported pregnancy or planning to become pregnant.
* Body weight greater than 300 pounds.
* Any condition in the opinion of the PI that would not allow safe conduct of study procedures (including IMR, MIP testing or step-test), such as a physical disability, recent musculoskeletal injury or illness, current and ongoing evaluation for undiagnosed cardiopulmonary or neurologic symptoms, undiagnosed chest pain, pneumothorax in the past 12 months, inner ear surgery in the past 12 months, or undiagnosed syncopal episodes.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2022-08-23 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Lang, MD, Principal Investigator — Duke University
Locations (1):
- Duke Healthy Lifestyles Clinic, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lang JE, Carrion VM, Bhammar DM, Howard JB, Armstrong SC. A Randomized Trial of Inspiratory Training in Children and Adolescents With Obesity. Child Obes. 2024 Oct;20(7):517-525. doi: 10.1089/chi.2023.0183. Epub 2024 May 2. PMID 38696657

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The Breathe-Fit trial was a single-center, partially-blinded, randomized 6-week parallel group intervention trial of inspiratory muscle training in youths with obesity being seen at the Duke Healthy Lifestyles childhood obesity treatment clinic. In brief, study staff screened the clinic schedule for initial eligibility and then approached potential patients to for recruitment and to confirm eligibility criteria and obtain consent/assent.
Period: Overall Study
Arm/Group | Active Inspiratory Muscle Rehabilitation (IMR) Group | SHAM
Started | 14 | 13
Completed | 12 | 13
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Inspiratory Muscle Rehabilitation (IMR) Group | SHAM | Total
Number analyzed (Participants) | 14 | 13 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.1 (2.8) | 11.5 (2.2) | 11.3 (2.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 9
  Male | 8 | 10 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 8
  Not Hispanic or Latino | 11 | 8 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 10 | 19
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14 | 13 | 27

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Complete Study Visit 3
Time Frame: approximately 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Active Inspiratory Muscle Rehabilitation (IMR) Group | SHAM
Number analyzed (Participants) | 14 | 13
Participants | 12 | 13

2. Primary Outcome: Adherence to Active IMR (Inspiratory Muscle Rehabilitation)
Description: Percentage of IMR completion (actual / planned reps over intervention period x 100)
Time Frame: up to 2 months
Measure: Median (Inter-Quartile Range); unit: percentage of completed repetitions
Arm/Group | Active Inspiratory Muscle Rehabilitation (IMR) Group | SHAM
Number analyzed (Participants) | 14 | 13
percentage of completed repetitions | 76 [55 to 96] | 69 [68 to 93]
Statistical Analysis 1: Comparison: Active Inspiratory Muscle Rehabilitation (IMR) Group vs SHAM; Repetition adherence; Test type: Other; p = 0.333, Chi-squared
Statistical Analysis 2: Comparison: Active Inspiratory Muscle Rehabilitation (IMR) Group vs SHAM; Session adherence; Test type: Other; p = 0.626, Chi-squared

3. Primary Outcome: Participant Satisfaction With IMR (Inspiratory Muscle Rehabilitation)
Description: Scored on a 5-point Likert scale where 1 = strongly disagree, 2 = disagree, 3 = neutral, 4 = agree, 5 = strongly agree.
Time Frame: up to 2 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Active Inspiratory Muscle Rehabilitation (IMR) Group | SHAM
Number analyzed (Participants) | 14 | 13
score on a scale | 5 [4.5 to 5] | 5 [4 to 5]
Statistical Analysis 1: Comparison: Active Inspiratory Muscle Rehabilitation (IMR) Group; Test type: Superiority; p = 0.416, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Change in Maximum Inspiratory Pressure (MIP) Over Intervention Period
Time Frame: Baseline, approximately 2 months
Measure: Mean (Standard Deviation); unit: cm water
Arm/Group | Active Inspiratory Muscle Rehabilitation (IMR) Group | SHAM
Number analyzed (Participants) | 14 | 13
cm water | 14 (37) | 7 (29)
Statistical Analysis 1: Comparison: Active Inspiratory Muscle Rehabilitation (IMR) Group vs SHAM; Test type: Superiority; p = 0.581, t-test, 2 sided

5. Secondary Outcome: Change in Modified Medical Research Council (mMRC) Dyspnea Scores Over Intervention Period
Description: The mMRC scale is a self-rating tool to measure the degree of disability that breathlessness poses on day-to-day activities on a scale from 0 to 4: 0, no breathlessness except on strenuous exercise; 1, shortness of breath when hurrying on the level or walking up a slight hill; 2, walks slower than people of same age on the level because of breathlessness or has to stop to catch breath when walking at their own pace on the level; 3, stops for breath after walking ∼100 m or after few minutes on the level; and 4, too breathless to leave the house, or breathless when dressing or undressing.
Time Frame: Baseline, approximately 2 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Inspiratory Muscle Rehabilitation (IMR) Group | SHAM
Number analyzed (Participants) | 14 | 13
score on a scale | -2.2 (1.5) | -1.1 (1.3)
Statistical Analysis 1: Comparison: Active Inspiratory Muscle Rehabilitation (IMR) Group vs SHAM; Test type: Superiority; p = 0.071, t-test, 2 sided

6. Secondary Outcome: Change in Average Daily Moderate-vigorous Physical Activity (MVPA) Time
Time Frame: Baseline, approximately 2 months
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | Active Inspiratory Muscle Rehabilitation (IMR) Group | SHAM
Number analyzed (Participants) | 14 | 13
minutes per day | 7 (15.7) | -16 (85)
Statistical Analysis 1: Comparison: Active Inspiratory Muscle Rehabilitation (IMR) Group vs SHAM; Test type: Superiority; p = 0.356, t-test, 2 sided

7. Secondary Outcome: Change in Average Daily Sedentary Physical Activity (SPA) Time
Description: Determined by the difference in MVPA between the baseline (run-in) value and value taken at the end of the intervention period.
Time Frame: Baseline, approximately 2 months
Population: Data not collected.
Arm/Group | Active Inspiratory Muscle Rehabilitation (IMR) Group | SHAM
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change in Average Daily Step Count
Time Frame: Baseline, approximately 2 months
Measure: Mean (Standard Deviation); unit: steps per day
Arm/Group | Active Inspiratory Muscle Rehabilitation (IMR) Group | SHAM
Number analyzed (Participants) | 14 | 13
steps per day | 865 (1134) | -51 (1341)
Statistical Analysis 1: Comparison: Active Inspiratory Muscle Rehabilitation (IMR) Group vs SHAM; Test type: Superiority; p = 0.079, t-test, 2 sided

9. Other Pre Specified Outcome: Heart Rate Change During 3-minute Step Test (HRC)
Description: determined by the change in HRC from baseline to final visit after intervention
Time Frame: Baseline, approximately 2 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Approximately 2 months
Arm/Group | Active Inspiratory Muscle Rehabilitation (IMR) Group | SHAM
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/13
Other Adverse Events (participants affected / at risk) | 0/14 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-26): https://cdn.clinicaltrials.gov/large-docs/34/NCT05412134/Prot_SAP_000.pdf